CLINICAL TRIAL: NCT01992367
Title: A Phase 1, Randomised, Double Blind, Placebo Controlled, 2-Part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Ascending Doses and Multiple Ascending Doses of ASLAN003 in Healthy Subjects
Brief Title: Phase 1, Randomised Double Blinded Placebo Controlled Study of ASLAN003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ASLAN003-001
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo arm
  Interventions: Drug: ASLAN003 ACTIVE
- ASLAN003 (Other): Active drug
  Interventions: Drug: ASLAN003 ACTIVE

INTERVENTIONS:
Drug: ASLAN003 ACTIVE — This is a single-centre, placebo-controlled, randomised, double-blind study involving SAD and MAD of ASLAN003 in healthy subjects.
  Other Names: ASLAN 003 , LAS186323

SUMMARY:
This is a single-centre, placebo-controlled, randomised, double-blind study to evaluate the safety and tolerability of single ascending doses (SAD) and multiple ascending doses (MAD) of ASLAN003 in healthy subjects

DETAILED DESCRIPTION:
This is a single-centre, placebo-controlled, randomised, double-blind study involving SAD and MAD of ASLAN003 in healthy subjects.

The study is divided into two parts:

* Part A: SAD cohorts and 1 cohort to assess food effect of ASLAN003 PK.
* Part B: MAD cohorts with one cohort being of healthy elderly subjects.

There will be a sentinel pair of subjects for each of SAD Cohorts 1, 2 and 3 who will be dosed first and then the same dose will be given to the rest of the subjects in the respective cohorts.

In addition, 8 subjects will receive ASLAN003 under both fed and fasted conditions

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for all subjects are as follows:
* are capable of understanding and complying with the requirements of the study and have signed the informed consent form (ICF);
* are able to communicate well with the Investigator, and understand and comply with the requirements of the study;
* male subjects aged between 21 and 50 years, inclusive (Part A and Cohorts 5, 6 and 7 of Part B only); male subjects and female subjects of non childbearing potential aged ≥55 years (Cohort 8 of Part B only);
* body mass index (BMI) in the range of 18 to 30 kg/m2, inclusive;
* healthy, as determined by pre study medical history, physical examinations, vital sign measurements, electrocardiogram (ECG; 12 lead reporting RR, PR, QRS, corrected QT [QTc] and QT interval corrected for heart rate using Fridericia's formulas [QTcF]) recordings with no evidence of clinically relevant medical disorders based on the opinion of the Investigator;
* whose out-of-normal range clinical laboratory test results are not clinically relevant and are acceptable to the Investigator;
* male subjects must be willing to use barrier contraception during sexual intercourse, i.e. condoms, even if their partners are post-menopausal, surgically sterile or are using accepted contraceptive methods, from the first day of dose administrations until 3 months after the last dose administration;

Exclusion Criteria:

* The exclusion criteria for all subjects are as follows:
* have participated in a study involving another investigational device or drug study within 90 days prior to randomisation in this study;
* history of drug hypersensitivity reactions or hypersensitivity to drugs chemically related to the IP;
* history or evidence of a clinically significant disorder, condition or disease (including, but not limited to, cardiopulmonary, oncologic, autoimmune, immunogenic, renal, metabolic, haematological or psychiatric), that, in the opinion of the Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion;
* existence of any surgical or medical condition which, in the judgement of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the IP;
* clinically significant history or evidence of any active or suspected bacterial, viral, fungal or parasitic infection within the 30 days prior to randomisation (e.g. common cold, viral syndrome, flu-like symptoms, etc.);
* active or recent history (within 30 days prior to randomisation) of acute viral infection of the skin (e.g. Herpes simplex, Molluscum contagiosum);
* active or history of psoriasis, or a first-degree relative with active or history of psoriasis;
* known history or evidence of active or latent tuberculosis infection (e.g. positive tuberculin skin test showing induration >5 mm or positive tuberculin blood test) in absence of previous Bacillus Calmette Guerin vaccination, or recent exposure (within 6 months prior to randomisation in this study) to an individual with active tuberculosis or with intention to travel to a country with a high risk of tuberculosis during the study period (including the follow up period);
* history of autoimmune disease including but not limited to lupus, rheumatoid arthritis, autoimmune thyroid disease and immune thrombocytopenia;
* with QT or QTcF values higher than 450 ms at screening;
* history of regular alcohol consumption (within 6 months prior to randomisation in this study), defined as: an average weekly intake of greater than 21 units or any average daily intake of greater than 3 units. One unit is equivalent to a half pint (220 mL) of beer or 1 (25 mL) measure of spirits or 1 glass (125 mL) of wine;

Ages: 21 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Safety | 6 months
  Safety assessments will include 12 lead ECGs, physical examiniation, vital signs measurements, pulse rate, RR, body temperature, clinical laboratory assessments and recording of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Please contact ASLAN Pharmaceuticals Pte Ltd, Study Director — contact@aslanpharma.com
Locations (1):
- Singapore, Singapore